CLINICAL TRIAL: NCT07325604
Title: Effect of Neuromuscular Electrical Stimulation on Unilaterial Central Facial Palsy: An Assesorblinded Randomized Controlled Trial
Brief Title: Effect of Neuromuscular Electrical Stimulation on Unilateral Central Facial Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Association of Occupational Therapist (Other); Hammel Neurorehabilitation Centre and University Research Clinic (Other); Hospital of Central Denmark Region, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 955087; 2501205 (Other: Medical Research Ethics Committees)
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Facial Palsy; Stroke
Keywords: NMES; Central facial palsy; Multicenter RCT; Stroke; Facial symmetry
MeSH Terms: conditions — Facial Paralysis; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NMES (Experimental): NMES is provided as an add-on to usual care
  Interventions: Device: Neuromuscular electrical stimulation (NMES); Other: Usual Care
- Usual care (Active Comparator): This arm receives usual care of facial palsy without NMES. Usual care encompass mimical exercises, facio oral sensory input, and kinesio taping.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — Electrical stimulation of facial muscles.
  Arms: NMES
Other: Usual Care — This arm receives usual care of facial palsy without NMES. Usual care encompass mimical exercises, facio oral sensory input, and kinesio taping.

SUMMARY:
Background Central facial palsy (CFP) is a common condition in stroke, with an estimated prevalence of 45%. CFP can lead to facial asymmetry, problems with mouth closure and food processing, bite marks on the cheek, social isolation, and reduced quality of life. CFP is seen as an important area of rehabilitation, and training is therefore often carried out to reduce the consequences of CFP. In a recent systematic review conducted by the principal investigator, the results showed that very few studies have been conducted that have investigated the effect of training for CFP, and there is currently no scientific evidence to support the effect of the various training interventions.

Objective To investigate the effect of Neuromuscular electrical stimulation (NMES) on facial symmetry compared to usual practice, in participants with CFP as a result of stroke.

Hypothesis: Participants who receive training with NMES together with usual training for facial paralysis have greater improvement in facial symmetry than participants who only receive usual training for facial paralysis.

Trial design Randomized controlled trial (RCT) with a nested pilot trial. A pilot trial/RCT will be conducted in order to power calculation in an RCT. The protocol for the pilot trial and RCT will be the same, and participants from the pilot trial and their outcome data are thus expected to be included in the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Central facial palsy
* First time stroke
* >=18 years
* Able to provide written consent

Exclusion Criteria:

* Not able to cooperate for mimical exercises
* Contraindications for NMES
* Admitted for three weeks assessment stay at the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
My Facial Quantification (MyFacialQ) | From enrollment to the end of treatment at four weeks"
  MyFacialQ quantifies degree of unilateral facial palsy through video recordings of mimical exercises. The development and validation study for MyFacialQ is in review.

SECONDARY OUTCOMES:
Iowa Oral Performance Instrument (IOPI) | From enrollment to the end of treatment at four weeks
  Measurement of lip strength
Facial Clinimetric Evaluation (FACE) | From enrollment to three months follow-up after the intervention
  Patient reported outcome on facial palsy

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Fabricius, PhD, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic & Department of clinical medicine, Aarhus University
Locations (1):
- Hammel neurorehabilitation centre and university research clinic, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD raw data is mainly video recordings, and these will not be shared. However aggregated measures from the video recordings may be shared.